CLINICAL TRIAL: NCT02127684
Title: Frequent Dosing Regimen of Lucentis for Subjects With Persistent Diabetic Macular Edema Despite Standard AntiVEGF Dosing
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor determined study design would not produce useful results
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML29381
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Persistent Diabetic Macular Edema
Keywords: diabetic macular edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Dosing Group (Active Comparator): Standard Dosing Group will receive intravitreal injections of 0.3mg. ranibizumab at baseline, week 4 and 8 )sham injections at week 2 and 6). After week 8 retreatment will be given monthly if edema is greater than 290um or ETDRS visual acuity score <83
  Interventions: Drug: ranibizumab
- Frequent dosing group (Experimental): Frequent dosing subjects will be evaluated and treated every two weeks through week 8 with intravitreal injection of 0.3mg ranibizumab. Subjects will then be evaluated monthly through week 24 and will receive treatment with ranibiumab based on residual edema and visual acuity
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — ranibizumab 0.3mg intravitreally monthly
  Other Names: Lucentis
  Arms: Standard Dosing Group
Drug: ranibizumab — ranibizumab given every 2 weeks for 8 weeks then monthly as needed
  Other Names: Lucentis
  Arms: Frequent dosing group

SUMMARY:
The investigators would like to investigate the efficacy of more frequent treatment with Lucentis for subjects with persistent diabetic macular edema despite standard dosing regimen.

DETAILED DESCRIPTION:
This is an open-label, subject masked, phase II study of intravitreally administered ranibizumab in subjects with persistent diabetic macular edema. Persistent diabetic macular edema is defined as subjects who still have central subfield thickness on SD-OCT of greater than 320 microns after having received at least 3 previous doses of AntiVEGF therapy in the past 5 months. Consented, enrolled subjects will be randomized into two subgroups: (1) standard dosing of monthly 0.3mg ranibizumab or (2) 0.3mg ranibizumab given 2 weeks apart for 5 doses followed by monthly dosing.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age >18 years
* Diagnosis of Type 1 or Type 2 diabetes
* BCVA score using the ETDRS method of >24 and <78 in the study eye at the screening visit
* 3 or more intravitreal injections of AntiVEGF over the 5 months prior to screening
* Presence of diabetic macular edema defined as SD-OCT CST >320 microns on spectral domain machine

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  * Anti-VEGF treatment in the study eye within 3 weeks prior to screening
  * Intravitreal Ozurdex treatment in the study eye within 12 weeks prior to screening
  * Intravitreal steroid treatment in the study eye within 8 weeks prior to screening
  * PRP or focal laser in the study eye within 4 months prior to screening
  * Active iris neovascularization in the study eye
  * Any ocular condition in the study eye that, in the opinion of the investigator, is severe enough to compromise the study result.
  * History of cataract surgery in the study eye within 3 months prior to screening visit
  * Uncontrolled systemic disease
  * Current enrollment in an investigational drug study or participation in such a study within 30 days prior to the screening visit
  * Female patients who are pregnant, nursing or planning a pregnancy or who are of childbearing potential and not using a reliable means of contraception.
  * Any condition or reason (including inability to read ETDRS chart or language barrier) that precludes the patient's ability to comply with study requirements including completion of the study.
  * Known allergy, hypersensitivity or contraindication to the study medications, its components, fluorescein or povidone iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
mean change in optical coherence topography central subfield thickness at 12 weeks and 24 weeks after randomization | 24 weeks
  mean change in optical coherence topography central subfield thickness at 12 weeks and 24 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Raj K. maturi MD PC
Locations (1):
- Raj K Maturi MD, Indianapolis, Indiana, United States